CLINICAL TRIAL: NCT02643849
Title: Use of The Spanner® Temporary Prostatic Stent as an Alternative to a Urinary Catheter to Achieve Bladder Drainage in Men Unfit for Other Treatments
Brief Title: Use of The Spanner Temporary Prostatic Stent as an Alternative to a Urinary Catheter to Achieve Bladder Drainage in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SRS Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRS 1.0
Record Dates: First submitted 2015-12-22; First posted 2015-12-31 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spanner (Experimental)
  Interventions: Device: The Spanner Temporary Prostatic Stent

INTERVENTIONS:
Device: The Spanner Temporary Prostatic Stent

SUMMARY:
The Spanner is being evaluated for use to manage voiding dysfunction and lower urinary tract symptoms in subjects to achieve bladder drainage in men unfit for other treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age > 45 years;
* In urinary retention and catheterized (indwelling or intermittent) for less than 180 days;
* Documented diagnostic history (within 180 days of study) of detrusor contractility (>= 15 cmH2O) confirmed via pressure-flow test;
* Negative Urinalysis on Visit 1;
* Not a candidate for pharmacologic, minimally invasive or surgical treatment of the prostate;
* Charlson Weighted Index of Comorbidity Score >= 1;
* Willing and able to sign the Informed Consent Form;
* Willing and able to complete the follow-up protocol requirements;
* Experiencing catheter-induced discomfort.

Exclusion Criteria:

* Current use of a urinary catheter daily for greater than 180 consecutive days immediately preceding entering into the study;
* Positive Urinalysis on Visit 1;
* Current or recent (within the last 6 months) urinary tract disease including urethral stricture, bladder stones, and other significant urological conditions or surgery;
* Surgery altering the normal uro-genital anatomy or abnormal urethral anatomy that affect the function of the lower urinary tract;
* History of conditions associated with neurogenic bladder, including spinal cord injury, multiple sclerosis, or Parkinson's disease;
* Use of anticholinergic medication;
* Gross hematuria when catheter is removed on Visit 1;
* Known or suspected prostate cancer;
* Prior pelvic irradiation therapy;
* Prostatic urethral length < 4 cm or > 9 cm (combined length from the top proximal side of the bladder neck to the bottom distal side of the external sphincter);
* Intravesical enlargement of the median lobe of the prostate.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Atlantic Urology, Daytona Beach, Florida
  - Advanced Urology Specialists, Oxford, Florida
  - Urology Specialists of West Florida, Palm Harbor, Florida
  - Pinellas Urology Inc, South Pasadena, Florida
  - Greater Boston Urology, Hingham, Massachusetts
  - Brooklyn Urology Research Group, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 109 subjects were screened for inclusion. Two subjects were excluded because they did not meet all inclusion/exclusion criteria and did not participate. Therefore the Intent to Treat population was 107 subjects, each of whom received at least 1 stent insertion.
Groups:
- Spanner: The Spanner Temporary Prostatic Stent
Period: Overall Study
Arm/Group | Spanner
Started | 107
Completed | 82
Not Completed | 25

BASELINE CHARACTERISTICS:
Population: All study subjects were catheter dependent, with comorbid conditions and were on medications/treatment regiments for those conditions.
Arm/Group | Spanner
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.12 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 104
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 107

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Post-void Residual (PVR) of ≤150 ml Over 90 Days
Description: To determine the percentage of subjects who achieved adequate bladder drainage over 90 days, defined as a PVR of ≤150 ml.
Time Frame: 90 days
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Spanner
Number analyzed (Participants) | 107
Participants | 79

2. Secondary Outcome: Number of Participants Who Achieved Post-void Residual (PVR) of ≤150 ml Over 30 Days
Description: To determine the percentage of subjects who achieved adequate bladder drainage over 30 days, defined as a PVR of ≤150 ml.
Time Frame: 30 days
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Spanner
Number analyzed (Participants) | 107
Participants | 86

3. Other Pre Specified Outcome: The Distribution of International Prostate Symptom Score (IPSS Score) Over 90 Days
Description: To determine the distribution of IPSS Scores at each stent replacement visit (Visit 2, 3 and 4). The IPSS Score is calculated from the responses to seven questions related to the severity and frequency of symptoms of benign prostatic hyperplasia (BPH). Each of the seven scored questions are put on a scale of 0-5, with the score of 5 being the worst score and the most severe symptom. The scores for the seven questions are added up and the IPSS score therefore ranges from 0-35, with 0 being the best score and 35 being the worst score. Scores of 0-7 are categorized as "Mild Symptoms". Scores of 8-19 are categorized as "Moderate Symptoms". Scores of 20-35 are categorized as "Severe Symptoms".
Time Frame: 30, 60 and 90 days
Population: All active patients in the Intent to Treat Population. On Visit 2, 89 subjects remained active in the study. On Visit 3 and Visit 4 82 subjects remained active in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spanner
Number analyzed (Participants) | 107
score on a scale
  Visit 2 (30 days): number analyzed (Participants) | 89
  Visit 2 (30 days) | 7.70 (6.84)
  Visit 3 (60 days): number analyzed (Participants) | 82
  Visit 3 (60 days) | 7.55 (6.24)
  Visit 4 (90 days): number analyzed (Participants) | 82
  Visit 4 (90 days) | 7.11 (6.1)

4. Other Pre Specified Outcome: The Average Maximum Flow Rate Over 90 Days
Description: To determine the average and standard deviation of QMax at each stent visit (Visits 1-4)
Time Frame: 1, 30, 60 and 90 days
Population: All active patients in the Intent to Treat Population who voided prior to the PVR measurement during each visit.
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Spanner
Number analyzed (Participants) | 107
ml/s
  Visit 1 (Day 1): number analyzed (Participants) | 93
  Visit 1 (Day 1) | 11.91 (6.95)
  Visit 2 (30 days): number analyzed (Participants) | 84
  Visit 2 (30 days) | 11.37 (7.09)
  Visit 3 (60 days): number analyzed (Participants) | 73
  Visit 3 (60 days) | 11.77 (6.43)
  Visit 4 (90 days): number analyzed (Participants) | 73
  Visit 4 (90 days) | 9.55 (5.42)

ADVERSE EVENTS:
Time Frame: AE Data was collected from time of enrollment through 14 days after the final stent was removed, up to 4 months.
Arm/Group | Spanner
All-Cause Mortality (participants affected / at risk) | 0/107
Serious Adverse Events (participants affected / at risk) | 15/107
Other Adverse Events (participants affected / at risk) | 81/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spanner (N=107)
Abdominal pain (Gastrointestinal disorders) | 1
Weakness (General disorders) | 2
Clostridium difficile toxin test positive and E. coli urinary tract infection (Infections and infestations) | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 2
Flank discomfort and dysuria (General disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Intervertebral disc operation (Musculoskeletal and connective tissue disorders) | 1
Malignant and unspecified neoplasms gastrointestinal (Gastrointestinal disorders) | 1
Hypotension and dehydration (General disorders) | 1
Shortness of breath and fever (General disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Fever, flu and mental state abnormal (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Fatigue and fever (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spanner (N=107)
Bacteriuria (Renal and urinary disorders) | 25
Pain (General disorders) | 10
Urinary urgency (Renal and urinary disorders) | 8
Urinary frequency (Renal and urinary disorders) | 6
Dysuria (Renal and urinary disorders) | 6
Voiding difficulty (Renal and urinary disorders) | 6
Hematuria (Renal and urinary disorders) | 5
Urinary incontinence (Renal and urinary disorders) | 4
Urinary retention (Renal and urinary disorders) | 4
Urinary tract infection (Renal and urinary disorders) | 4
Penile pain (Renal and urinary disorders) | 3
Residual urine (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02643849/SAP_000.pdf
  • Study Protocol (2016-01-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT02643849/Prot_001.pdf